CLINICAL TRIAL: NCT05743218
Title: Clinical Study of Liver Meridian in the Treatment of Male Impotence and Female Premature Ovarian Failure
Brief Title: Clinical Efficacy of Acupuncture on the Liver Meridian in Women With Diminished Ovarian Reserve
Acronym: GJZLLCCBGNXJ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019YFC1709104-1
Record Dates: First submitted 2023-01-12; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Ovarian Reserve; Acupuncture Therapy; Meridian
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: The subjects were randomly assigned to the liver meridian group, the stomach meridian group and the non-acupoint acupuncture groups group at a ratio of 1:1:1.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: On account of the particularity of acupuncture research, it is impossible to blind acupuncture operators. Blinded evaluation will be adopted in the trial, and the third party who does not know the grouping will evaluate the efficacy. Blind statistical analysis was used in the data summary stage, and the researchers, operators and statisticians were separated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- liver meridian group (Experimental): Four acupoints; LR3 Taichong, LR5 Ligou, LR8 Ququan, and LR12 Jiman. Based on the national standard of the People's Republic of China in 2006 (GB/T 12346-2006). The patient will be in a supine position. Taichong will be punctured at a 25-mm depth using a 0.35×25-mm filiform needle, Ligou will be punctured at a 15-20-mm depth with a 0.35×25-mm filiform needle, Ququan at a 20-25-mm depth with a 0.30×40-mm filiform needle, and an acute pulse of 15-20 mm. Each acupoint will be subject to a small amount of uniform lifting and twisting to the degree of local acid distension. An auxiliary needle (0.16×13 mm) will be inserted approximately 5 mm into the needle, 2 mm proximal to the heart of each acupoint along the meridian. The negative electrode will be connected to the main point, and the positive electrode will be connected to the auxiliary needle, and connect the electroacupuncture instrument. The needles will be retained for 30 min respectively, once every other day, 36 treatments.
  Interventions: Other: electropuncture
- stomach meridian group (Active Comparator): Four acupoints have been selected for the gastric meridian group, including ST42 Chongyang, ST40 Fenglong, ST36 Zusanli, and ST31 Biguan. The acupoint locations are based on the national standard of the People's Republic of China in 2006 (GB/T 12346-2006). The patient will be supine during the procedure, and the needles will be routinely sterilized. Straight needling will be performed in the hip region using a 0.30×50-mm-filiform needle, a 0.30×50-mm filiform needle in Zusanli, and a 0.30×40-mm filiform needle in Fenglong. A 0.35×25-mm filiform needle will be used to stimulate Chongyang for 10-15 mm, and each acupoint will be gently and evenly lifted, inserted, and twisted to local acid distension. Electroacupuncture will be applied in the same manner as for the liver meridian group. The needles will be retained for 30 min respectively, once every other day, then thrice weekly for a total of 36 treatments in the three groups.
  Interventions: Other: electropuncture
- non-acupoint acupuncture group (Placebo Comparator): Four points: (1) On the lateral thigh, between the vastus lateralis and biceps femoris, the midpoint of the popliteal stria, and the highest point of the greater trochanter. (2) On the lateral side of the calf, beside the level of Zusanli, and at the lateral edge of the tibia. (3) On the fibular side of the calf, the midpoint of the stomach meridian, and the bile meridian, 3 cm above the tip of the lateral malleolus and in front of the hanging bell. (4) On the lateral side of the calcaneus, and the servant enters the midpoint of the line connecting the posterior edge of the calcaneus at the same level. The 0.30×25-mm filiform needles are inserted straight for 3-5 mm at the points, the needles can stand without Deqi. The auxiliary needle will be inserted and electroacupuncture will be connected (same as in the other group). The internal wire of the electroacupuncture instrument will be interrupted, no current passed through. The treatment time is the same as the other two groups.
  Interventions: Other: electropuncture

INTERVENTIONS:
Other: electropuncture — Electroacupuncture (EA) is a method of treating diseases by inserting a needle (usually a filiform needle) into the skin or tissue of a patient at a certain Angle, and then passing through the needle (sensing) micro-current waves of human bioelectricity to stimulate specific parts of the human body (acupoints).
  1. Disposable sterile acupuncture filiform needle (0.16mm×13mm, 0.30mm×25mm, 0.30mm× 40mm), Guizhou Andi Medical Equipment Co, LTD, Guizhou Food and Drug Supervision and Equipment Production Xu 20170011.
  2. Electroacupuncture apparatus: SDZ-Ⅱ electroacupuncture apparatus of Huatuo brand, Suzhou Medical Supplies Factory Co., LTD., Registration No. : 20172270675.
  Other Names: acupuncture

SUMMARY:
Diminished ovarian reserve (DOR) refers to a decrease in the number and quality of oocytes in the ovary, which results in impaired ovarian function and decreased fertility. Meanwhile, levels of the anti-Müllerian hormone (AMH), antral follicle count (AFC), and Follicle-Stimulating Hormone (FSH) also decrease in patients with DOR. In general, there is a decline in fertility and premature menopause. Some patients will have low menstrual volume, oligomenorrhea or even amenorrhea, abnormal uterine bleeding, ovulation disorders, infertility and perimenopausal performance before the age of 40, and eventually develop into premature ovarian failure. In recent years, with the changes of social culture, living environment, work pressure and other factors, the incidence of this disease has increased year by year, which has a great impact on women's fertility, mental health, quality of life, family relations and other aspects.

As a green and safe complementary and alternative therapy, acupuncture has been proved to be effective. According to the statistics, 904 (33.54%) of the 2695 syndromes indicated by acupoints of the liver meridian recorded in 93 ancient medical books are reproductive disorders, ranking first in the diseases indicated by the liver meridian and the 14 meridians. The body surface course of the liver meridian is closely related to the genitals, and there is a close relationship between the liver meridian and the genitals in physiology and pathology. According to the theory of the relationship between meridians and zangfu organs, the study aims to verify the efficacy and safety of acupuncture of the liver meridian and provide high-level research evidence for meridian syndrome differentiation of reproductive system diseases via "treatment from the liver."

DETAILED DESCRIPTION:
This is an exploratory multicenter randomized controlled trial involving four clinical research centers, including the First Affiliated Hospital of Hunan University of Traditional Chinese Medicine, Hubei Hospital of Traditional Chinese Medicine, Shaanxi Hospital of Traditional Chinese Medicine, and Guizhou Hospital of Traditional Chinese Medicine. Each clinical research center strictly screened cases according to the diagnostic criteria, inclusion criteria and exclusion criteria. After confirmation of enrollment, random numbers were obtained according to the application for random coding process until the total number of observation was completed. According to the sample size, a total of 198 patients with DOR need to be enrolled. The 29-week study period consists of a 4-week screening period, 1-week baseline period, 12-week treatment period, 12-week follow-up period, and assessments at baseline. He patients were randomly divided into three groups: the liver meridian, stomach meridian, and non-acupoint acupuncture groups. Due to the particularity of acupuncture research, it is impossible to blind acupuncture operators. Blinded evaluation will be adopted in the trial, and the third party who does not know the grouping will evaluate the efficacy. Blind statistical analysis was used in the data summary stage, and the researchers, operators and statisticians were separated. In the experimental group (liver meridian group), EA was applied to Taichong, Li gou, Ququan and Jimai. In the control group 1 (gastric meridian group), EA was applied to Chongyang, Fenglong, Zusanli and Biguan. In the control group 2 (the non-meridian non-acupoint group), 4 non-meridian non-acupoints were selected from the lateral thigh, the lateral calf and the lateral calcaneus, respectively (see the treatment methods of the non-meridian non-acupoint group for details) and stimulated with EA.

The main evaluation index will be Anti-Müllerian hormone(AMH), The secondary evaluation index include serum sex hormones (bFSH, bE2, bLH, bFSH/bLH), antral follicle count(AFC),, menstrual status, the modified Kupperman Index(KI), perimenopausal quality of life score (MENQOL) ,Self-Rating Anxiety Scale( SAS ), self-rating depression scale(SDS), Menstrual conditions. The patients were evaluated at different time points during the baseline period, treatment period and follow-up period, and the incidence of adverse events will be recorded. Double data entry will be used in this trial to ensure the accuracy of data entry. A three-level quality control system (self-inspection by each center, supervision by project management team, and third-party audit) was implemented to ensure that the implementation, recording and reporting of clinical trials were in accordance with the trial protocol, standard operating procedures, and relevant laws and regulations. The statistical analysis plan was developed by the statistical analysis principal and the principal investigators in accordance with the protocol and was finalized before the database was locked. The tables for the statistical analysis were developed. Statistical analysis will be calculated by SPSS25.0 statistical analysis software, P<0.05 (i.e., =0.05) will be considered statistically significant, in order to clarify the efficacy and safety of acupuncture on DOR.

ELIGIBILITY:
Inclusion Criteria:

- The inclusion criteria are as follows:

1. patients with the detection indicators within 3 months before enrollment met the diagnostic criteria of DOR.
2. patients aged between 18 and 40 years old.
3. patients who have received no other treatment in the 2 months before enrollment. (4) patients who voluntarily participate in this study and can actively cooperate with the study process.

(5) patients who have signed an informed consent form. Patients who meet all five criteria will be eligible for this study.

Exclusion Criteria:

* (1) Patients with polycystic ovarian syndrome, hyperprolactinemia, pituitary or hypothalamic amenorrhea, thyroid dysfunction, congenital malformations, and organic lesions in the reproductive organs.

  (2) Patients with a history of local ovarian surgery, such as oophorectomy and ovarian tumor surgery.

  (3) Patients with a history of chemotherapy or pelvic radiotherapy and a history of therapy with immunosuppressive agents.

  (4) Patients with comorbidities in the cardiovascular system, liver, kidney, hematopoietic system, nervous and mental system, diabetes, hypertension, and other diseases.

  (5) Patients being administered estrogen, progesterone, or dehydroepiandrosterone (DHEA) within 2 months before enrollment.

  (6) Patients who cannot tolerate blood or ultrasound testing. (vii) Patients who are also participating in other clinical trials.

  (7) Patients who refuse to sign the informed consent form. Patients who meet any of the above criteria will be excluded.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 198 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The value of anti-mullerian hormone(AMH) | 3 checkpoints. Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks) and enrollment 24 weeks(Changes at 12 weeks of treatment and 12 weeks of follow-up).
  This index is used to measure ovarian hormone secretion function and assess ovarian reserve function. Instrument:Beckman Coulter Access automatic immune analyzer.
  Method: Venous blood will be collected on an empty stomach at 3-5mL in the morning on the 2nd to 4th day of menstruation, centrifuged at 5000r/min for 3min with a high-speed centrifuge, and the upper serum is taken and stored in a -80℃ refrigerator for test.
  Unit: ng/mL.

SECONDARY OUTCOMES:
The number of antral follicle count (AFC) | 3 checkpoints. Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks) and enrollment 24 weeks(Changes at 12 weeks of treatment and 12 weeks of follow-up).
  The number of antral follicles was detected by three-dimensional B-ultrasound to evaluate ovarian reserve function. The smaller the number, the more severe the symptoms.
Sex hormone: follicle-stimulating hormone (FSH), luteinizing hormone (LH), estradiol (E2） | 3 checkpoints. Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks) and enrollment 24 weeks(Changes at 12 weeks of treatment and 12 weeks of follow-up).
  Use Chemiluminescence immunoassay to detected the ovarian hormone secretion. On the 2nd to 4th day of menstruation, 5 ml of venous blood will be collected from subjects in the morning under the condition of fasting for 8 h and put into the test tube without anticoagulant. The collected samples will be centrifuged to separate the upper serum and stored in the refrigerator at -70℃ for examination. Unit: FSH(mLU/mL), LH(mLU/mL), E2( pg/mL).
The total score of the modified Kupperman scale | 3 checkpoints. Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks) and enrollment 24 weeks(Changes at 12 weeks of treatment and 12 weeks of follow-up).
  To evaluate the severity of perimenopausal syndrome symptoms.Each item has a different basic and severity score, the severity score is calculated according to 0-3 points, and the symptom score is calculated as follows:Symptom score=basic score×severity score.The sum of each symptom score is the total score; the higher the total score, the more severe the disease. Patients with a normal score have <6 points. This with mild, moderate, and severe disease have 6-15, 16-30, and >30 points, respectively.
The total score of the perimenopausal quality of life score | 3 checkpoints. Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks) and enrollment 24 weeks(Changes at 12 weeks of treatment and 12 weeks of follow-up).
  29 items, divided into Vasomotor symptoms, psychosocial function, physical function, sexual life, each item scored 1-7 points.
  Dimension score = Total score of item questions in each dimension ➗ Number of questions Total score = Sum of four dimensions scores
The total score of the self-rating anxiety Scale | 3 checkpoints. Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks) and enrollment 24 weeks(Changes at 12 weeks of treatment and 12 weeks of follow-up).
  Reflect anxiety level. 20 items, each item 1-4 points, total score and standard score (total score ×1.25), the higher the score, the more severe symptoms.
The total score of the self-rating Depression Scale | 3 checkpoints. Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks) and enrollment 24 weeks(Changes at 12 weeks of treatment and 12 weeks of follow-up).
  Reflect the degree of depression. 20 items, each item 1-4 points, total score and standard score (total score ×1.25), the higher the score, the more severe symptoms.
Menstrual assessment | Enrollment 1、4、8、12、16、20、24 weeks.
  Menstruation was assessed throughout the study period (a total of 7 times). The evaluation consists of 6 items, each item is scored (0 to 4 points), and the total score is calculated for each time. The lower the total score is, the better the menstrual condition is.

OTHER OUTCOMES:
White blood cell (WBC) | Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks).
  Normal value (unit): 3.5-9.5 (109/L). Assessment with reference to the normal range. 1- Normal (Within the reference range) 2- Abnormal (Outside the reference range). The purpose is to evaluate whether acupuncture has an effect on WBC, which is a safety assessment.
Red blood cell (RBC) | Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks)
  Normal value (unit): 3.8-5.1(1012/L). Assessment with reference to the normal range. 1- Normal (Within the reference range) 2- Abnormal (Outside the reference range). The purpose is to evaluate whether acupuncture has an effect on RBC, which is a safety assessment.
Blood platelet | Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks)
  Normal value (unit): 125-350(109/L). Assessment with reference to the normal range. 1- Normal (Within the reference range) 2- Abnormal (Outside the reference range). The purpose is to evaluate whether acupuncture has an effect on Blood platelet, which is a safety assessment.
Hemoglobin | Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks)
  Normal value (unit): 115-150 (g/L). Assessment with reference to the normal range. 1- Normal (Within the reference range) 2- Abnormal (Outside the reference range). The purpose is to evaluate whether acupuncture has an effect on Hemoglobin, which is a safety assessment.
Alanine aminotransferase(ALT) | Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks)
  Normal value (unit): 0-33(IU/L). Assessment with reference to the normal range. 1- Normal (Within the reference range) 2- Abnormal (Outside the reference range). The purpose is to evaluate whether acupuncture has an effect on ALT, which is a safety assessment.
Aspartate aminotransferase (AST) | Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks)
  Normal value (unit): 0-32(IU/L). Assessment with reference to the normal range. 1- Normal (Within the reference range) 2- Abnormal (Outside the reference range). The purpose is to evaluate whether acupuncture has an effect on AST, which is a safety assessment.
Blood - urea nitrogen (UREA) | Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks)
  Normal value (unit): 2.14-7.14 (umol/L). Assessment with reference to the normal range. 1- Normal (Within the reference range) 2- Abnormal (Outside the reference range). The purpose is to evaluate whether acupuncture has an effect on UREA, which is a safety assessment.
Creatinine (CREA) | Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks)
  Normal value (unit): 45-84 (umol/L). Assessment with reference to the normal range. 1- Normal (Within the reference range) 2- Abnormal (Outside the reference range). The purpose is to evaluate whether acupuncture has an effect on CREA, which is a safety assessment.
Prothrombin time (PT) | Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks)
  Normal value (unit): 11-14(s). Assessment with reference to the normal range. 1- Normal (Within the reference range) 2- Abnormal (Outside the reference range). The purpose is to evaluate whether acupuncture has an effect on PT, which is a safety assessment.
Activated partial thromboplastin time(ATPP) | Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks)
  10.Activated partial thromboplastin time(ATPP)
Thrombin time(TT) | Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks)
  Normal value (unit): 20 (s). Assessment with reference to the normal range. 1- Normal (Within the reference range) 2- Abnormal (Outside the reference range). The purpose is to evaluate whether acupuncture has an effect on TT, which is a safety assessment.
Fibrinogen concentration(FBI) | Baseline period(1 week before enrollment), enrollment 12 weeks (Change from Baseline at 12weeks)
  Assessment with reference to the normal range. 1- Normal (Within the reference range) 2- Abnormal (Outside the reference range). The purpose is to evaluate whether acupuncture has an effect on FBI, which is a safety assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Hunan University of Chinese Medicine, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
ur subject database is called Zintuikang Integrated Big Data Application Platform, and other researchers can access it through the website. The administrator set up the account, and other researchers can log in by changing the password after registration. Their account has the authority to access the data and enter the CRF form.

REFERENCES:
- [Background] Practice Committee of the American Society for Reproductive Medicine. Electronic address: asrm@asrm.org; Practice Committee of the American Society for Reproductive Medicine. Testing and interpreting measures of ovarian reserve: a committee opinion. Fertil Steril. 2020 Dec;114(6):1151-1157. doi: 10.1016/j.fertnstert.2020.09.134. PMID 33280722
- [Background] Sun W, Stegmann BJ, Henne M, Catherino WH, Segars JH. A new approach to ovarian reserve testing. Fertil Steril. 2008 Dec;90(6):2196-202. doi: 10.1016/j.fertnstert.2007.10.080. Epub 2008 Apr 22. PMID 18433750
- [Background] Cohen J, Chabbert-Buffet N, Darai E. Diminished ovarian reserve, premature ovarian failure, poor ovarian responder--a plea for universal definitions. J Assist Reprod Genet. 2015 Dec;32(12):1709-12. doi: 10.1007/s10815-015-0595-y. Epub 2015 Oct 13. PMID 26463876
- [Background] Wang Y, Li Y, Chen R, Cui X, Yu J, Liu Z. Electroacupuncture for reproductive hormone levels in patients with diminished ovarian reserve: a prospective observational study. Acupunct Med. 2016 Oct;34(5):386-391. doi: 10.1136/acupmed-2015-011014. Epub 2016 May 13. PMID 27177929
- [Background] Atasever M, Soyman Z, Demirel E, Gencdal S, Kelekci S. Diminished ovarian reserve: is it a neglected cause in the assessment of recurrent miscarriage? A cohort study. Fertil Steril. 2016 May;105(5):1236-1240. doi: 10.1016/j.fertnstert.2016.01.001. Epub 2016 Jan 21. PMID 26806685
- [Background] Steiner AZ, Pritchard D, Stanczyk FZ, Kesner JS, Meadows JW, Herring AH, Baird DD. Association Between Biomarkers of Ovarian Reserve and Infertility Among Older Women of Reproductive Age. JAMA. 2017 Oct 10;318(14):1367-1376. doi: 10.1001/jama.2017.14588. PMID 29049585
- [Background] Bunnewell SJ, Honess ER, Karia AM, Keay SD, Al Wattar BH, Quenby S. Diminished ovarian reserve in recurrent pregnancy loss: a systematic review and meta-analysis. Fertil Steril. 2020 Apr;113(4):818-827.e3. doi: 10.1016/j.fertnstert.2019.11.014. Epub 2020 Mar 4. PMID 32145928
- [Background] Birch S, Lee MS, Kim TH, Alraek T. On defining acupuncture and its techniques: A commentary on the problem of sham. Integr Med Res. 2022 Jun;11(2):100834. doi: 10.1016/j.imr.2022.100834. Epub 2022 Jan 8. No abstract available. PMID 35111572
- [Background] Hong L, Peng S, Li Y, Fang Y, Wang Q, Klausen C, Yin C, Wang S, Leung PCK, Yang X. miR-106a Increases Granulosa Cell Viability and Is Downregulated in Women With Diminished Ovarian Reserve. J Clin Endocrinol Metab. 2018 Jun 1;103(6):2157-2166. doi: 10.1210/jc.2017-02344. PMID 29590425
- [Background] Maioli C, Falciati L, Marangon M, Perini S, Losio A. Short- and long-term modulation of upper limb motor-evoked potentials induced by acupuncture. Eur J Neurosci. 2006 Apr;23(7):1931-8. doi: 10.1111/j.1460-9568.2006.04698.x. PMID 16623849
- [Background] Zhao L, Chen J, Li Y, Sun X, Chang X, Zheng H, Gong B, Huang Y, Yang M, Wu X, Li X, Liang F. The Long-term Effect of Acupuncture for Migraine Prophylaxis: A Randomized Clinical Trial. JAMA Intern Med. 2017 Apr 1;177(4):508-515. doi: 10.1001/jamainternmed.2016.9378. PMID 28241154
- [Background] Liu CZ, Xie JP, Wang LP, Liu YQ, Song JS, Chen YY, Shi GX, Zhou W, Gao SZ, Li SL, Xing JM, Ma LX, Wang YX, Zhu J, Liu JP. A randomized controlled trial of single point acupuncture in primary dysmenorrhea. Pain Med. 2014 Jun;15(6):910-20. doi: 10.1111/pme.12392. Epub 2014 Mar 17. PMID 24636695
- [Background] Brinkhaus B, Hummelsberger J, Kohnen R, Seufert J, Hempen CH, Leonhardy H, Nogel R, Joos S, Hahn E, Schuppan D. Acupuncture and Chinese herbal medicine in the treatment of patients with seasonal allergic rhinitis: a randomized-controlled clinical trial. Allergy. 2004 Sep;59(9):953-60. doi: 10.1111/j.1398-9995.2004.00540.x. PMID 15291903
- [Background] di Clemente N, Racine C, Pierre A, Taieb J. Anti-Mullerian Hormone in Female Reproduction. Endocr Rev. 2021 Nov 16;42(6):753-782. doi: 10.1210/endrev/bnab012. PMID 33851994
- [Background] Sun XY, Lan YZ, Liu S, Long XP, Mao XG, Liu L. Relationship Between Anti-Mullerian Hormone and In Vitro Fertilization-Embryo Transfer in Clinical Pregnancy. Front Endocrinol (Lausanne). 2020 Dec 4;11:595448. doi: 10.3389/fendo.2020.595448. eCollection 2020. PMID 33343511
- [Background] Hilditch JR, Lewis J, Peter A, van Maris B, Ross A, Franssen E, Guyatt GH, Norton PG, Dunn E. A menopause-specific quality of life questionnaire: development and psychometric properties. Maturitas. 1996 Jul;24(3):161-75. doi: 10.1016/s0378-5122(96)82006-8. PMID 8844630
- [Background] Zung WW. A rating instrument for anxiety disorders. Psychosomatics. 1971 Nov-Dec;12(6):371-9. doi: 10.1016/S0033-3182(71)71479-0. No abstract available. PMID 5172928
- [Background] Liu L, Pang R, Sun W, Wu M, Qu P, Lu C, Wang L. Functional social support, psychological capital, and depressive and anxiety symptoms among people living with HIV/AIDS employed full-time. BMC Psychiatry. 2013 Dec 1;13:324. doi: 10.1186/1471-244X-13-324. PMID 24289721